CLINICAL TRIAL: NCT04523623
Title: Oxycodone or Ibuprofen for Suspected Isolated Forearm Fractures in Pediatric Patients: A Randomized Noninferiority Trial
Brief Title: Pain Control Differences Between Oxycodone and Ibuprofen in Children With Isolated Forearm Injuries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project canceled for other reason , describe: - Lack of enrollment Project canceled - lack of enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OxyvsIbup2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Forearm Injuries; Pain, Acute; Pediatric ALL
Keywords: oxycodone; ibuprofen
MeSH Terms: conditions — Forearm Injuries; Acute Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Oxycodone; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen Group (Experimental): To compare analgesia from ibuprofen to oxycodone in the initial treatment of acute pain in suspected isolated forearm fractures in children.
  Interventions: Drug: Ibuprofen
- Oxycodone Group (Experimental): To compare analgesia from ibuprofen to oxycodone in the initial treatment of acute pain in suspected isolated forearm fractures in children.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — oxycodone 0.2mg/kg, max 10mg to be administered, randomized between that and Ibuprofen
  Arms: Oxycodone Group
Drug: Ibuprofen — ibuprofen 10mg/kg, max 800mg, randomized between that and Oxycodone
  Arms: Ibuprofen Group

SUMMARY:
Children presenting to the Emergency Room with the chief complaint of forearm injury and/or pain will be randomized to receive oral Oxycodone or Ibuprofen to control pain.

DETAILED DESCRIPTION:
A randomized, blinded cohort study. Consented patients will be randomized to receive either ibuprofen or oxycodone after initial RN patient assessment in Emergency Department Triage determines a need for radiographs to evaluate for possible forearm fracture. Pain assessment scores will be determined at Triage and at 30-minute intervals throughout the patient's course until the patient is discharged home or additional analgesic medication is administered.

ELIGIBILITY:
Inclusion Criteria:

1. 6 to 17 year old children presenting for care in the St. Louis Children's Hospital Emergency Department
2. Suspected acute (within 24 hours) isolated forearm fracture at the time of initial Triage assessment
3. American Society of Anesthesiologist physical status (ASA-PS) classification of I or II
4. Child with parent or legal guardian.

Exclusion Criteria:

1. Multiple injuries
2. Known adverse reaction to either ibuprofen or oxycodone pts with abnormal bones or metabolic conditions that affect bones
3. Administration of any opioid within 2 hours prior to presentation
4. Non-English speaking
5. Foster care, police custody, presenting without legal guardian

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Pain change/difference | 180 minutes total
  An appreciable change in pain scores (by 2 points) from presentation to discharge

REFERENCES:
- [Background] Ibuprofen or oxycodone? An observational cohort study of post emergency department discharge management of children's fracture pain. Ali S., Drendel A.L., Rosychuk R.J., Le May S., McGrath P., Carleton B., Johnson D.W. Canadian Journal of Emergency Medicine 2016 18 Supplement 1 (S47).
- [Background] Charney RL, Yan Y, Schootman M, Kennedy RM, Luhmann JD. Oxycodone versus codeine for triage pain in children with suspected forearm fracture: a randomized controlled trial. Pediatr Emerg Care. 2008 Sep;24(9):595-600. doi: 10.1097/PEC.0b013e3181850ca3. PMID 18772726
- [Background] Kircher J, Drendel AL, Newton AS, Dulai S, Vandermeer B, Ali S. Pediatric musculoskeletal pain in the emergency department: a medical record review of practice variation. CJEM. 2014 Nov;16(6):449-57. doi: 10.1017/s1481803500003468. PMID 25358276
- [Background] Chang AK, Bijur PE, Esses D, Barnaby DP, Baer J. Effect of a Single Dose of Oral Opioid and Nonopioid Analgesics on Acute Extremity Pain in the Emergency Department: A Randomized Clinical Trial. JAMA. 2017 Nov 7;318(17):1661-1667. doi: 10.1001/jama.2017.16190. PMID 29114833
- [Background] Ilyas AM, Miller AJ, Graham JG, Matzon JL. A Prospective, Randomized, Double-Blinded Trial Comparing Acetaminophen, Ibuprofen, and Oxycodone for Pain Management After Hand Surgery. Orthopedics. 2019 Mar 1;42(2):110-115. doi: 10.3928/01477447-20190221-02. Epub 2019 Feb 27. PMID 30810754
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Moradi M, Esmaeili S, Shoar S, Safari S. Use of oxycodone in pain management. Anesth Pain Med. 2012 Spring;1(4):262-4. doi: 10.5812/aapm.4529. Epub 2012 Apr 1. PMID 24904812
- [Background] Tsze DS, von Baeyer CL, Pahalyants V, Dayan PS. Validity and Reliability of the Verbal Numerical Rating Scale for Children Aged 4 to 17 Years With Acute Pain. Ann Emerg Med. 2018 Jun;71(6):691-702.e3. doi: 10.1016/j.annemergmed.2017.09.009. Epub 2017 Nov 6. PMID 29107409